CLINICAL TRIAL: NCT07066098
Title: A Multicenter, Randomized, Double-Blind, Phase III Study of IBI343 Monotherapy Plus Best Supportive Care Versus Placebo Plus Best Supportive Care in Participants With Claudin (CLDN) 18.2-Positive, Locally Advanced Unresectable or Metastatic Pancreatic Cancer Who Received>=2 Prior Lines of Therapy
Brief Title: A Multicenter Study of IBI343 Monotherapy Versus Placebo in Subjects With Previously Treated, Claudin (CLDN) 18.2-positive, Pancreatic Cancer(G-HOPE-002)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI343B302
Record Dates: First submitted 2025-06-26; First posted 2025-07-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): IBI343
  Interventions: Drug: IBI343
- Control Arm (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IBI343 — Subjects in the experimental arm will receive IBI343 6mg/kg intravenous infusion (IV) D1, Q3W in 3-week cycle
  Arms: Experimental Arm
Drug: Placebo — Subjects in the control arm will receive placebo 6mg/kg intravenous infusion (IV) D1, Q3W in 3-week cycle
  Arms: Control Arm

SUMMARY:
This is a study of a Multicenter, Randomized, Double-Blind, Phase III Study of IBI343 Monotherapy Plus Best Supportive Care Versus Placebo Plus Best Supportive Care in Participants with Claudin (CLDN) 18.2-Positive, Locally Advanced Unresectable or Metastatic Pancreatic Cancer Who Received at least 2 Prior Lines of Therapy. The primary objective of this study is to determine Overall Survival (OS) of IBI343 plus best supportive care (BSC) compared with placebo plus BSC.

DETAILED DESCRIPTION:
This is a study of a Multicenter, Randomized, Double-Blind, Phase III Study of IBI343 Monotherapy Plus Best Supportive Care Versus Placebo Plus Best Supportive Care in Participants with Claudin (CLDN) 18.2-Positive, Locally Advanced Unresectable or Metastatic Pancreatic Cancer Who Received at least 2 Prior Lines of Therapy. It is planned to enroll 201 participants, and participants will be randomized to receive IBI343 plus BSC or placebo plus BSC in a 2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the written informed consent form (ICF) and be willing and able to comply with the visits and related procedures stipulated in the plan.
2. Histologically confirmed unresectable locally advanced, or metastatic pancreatic cancer.
3. Have received and progression after at least two systemic therapies(must including a fluorouracil-based and a gemcitabine-based therapy).
4. ECOG PS score of 0 or 2.
5. Adequate bone marrow and organ function
6. Confirmed as CLDN18.2 positive.

Exclusion Criteria:

1. Participation in another interventional study, except observational or post-intervention follow-up.
2. Prior treatment with topoisomerase inhibitor-based ADC.
3. Has received the last dose of an anti-cancer therapy within 2 weeks or 5 half-lives (whichever is shorter) prior to the first dose of study treatment.
4. Plans to receive other anti-tumor treatments during treatment with the study drug (palliative radiotherapy for symptomatic (e.g., pain) relief that does not affect response assessment is allowed) .
5. Symptomatic CNS metastasis; asymptomatic brain metastases may be allowed with specific criteria.
6. History of other primary malignancies, except cured or low-risk of recurrence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
overall survival(OS) | approximately 24 months
  Overall survival (OS) is defined as the time from randomization to death from any cause.

SECONDARY OUTCOMES:
progression free survival(PFS) | approximately 24 months
  Progression-free survival (PFS) is defined as the time from random assignment in the trial to disease progression or death from any cause.
Objective response rate (ORR) | approximately 24 months
  ORR is defined as the proportion of subjects in the analysis population who achieve confirmed objective response (CR or PR) per RECIST v1.1.
disease control rate (DCR) | approximately 24 months
  DCR is defined as the proportion of subjects in the analysis population who achieve disease control (CR, PR, or SD) per RECIST v1.1 criteria.
duration of response (DoR) | approximately 24 months
  DoR is defined as the time from the first CR or PR to disease progression or death from any cause, whichever occurs first for subjects with ORR per RECIST v1.1 criteria.
time to response (TTR) | approximately 24 months
  TTR is defined as the time from randomization to the first CR or PR for subjects with ORR as assessed by IRRC per RECIST v1.1 criteria.
Adverse Event | approximately 24 months
  Adverse events will be assessed by investigator(s) according to NCI-CTCAE v5.0.
Area under the plasma concentration versus time curve (AUC) | approximately 24 months
  area under the curve (AUC) of single and multiple doses of IBI343
immunogenicity | approximately 24 months
  anti-drug antibody and/or neutralizing antibody
maximum concentration (Cmax) | approximately 24 months
  maximum concentration (Cmax) of single and multiple doses of IBI343
time to maximum concentration (Tmax) | approximately 24 months
  time to maximum concentration (Tmax) of single and multiple doses of IBI343

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China